CLINICAL TRIAL: NCT01386658
Title: A Multicenter, Open-Label, Non-Randomized Study to Assess the Pharmacokinetics, Tolerability, and Safety of a Single Subcutaneous Administration of Icatibant in Children and Adolescents With Hereditary Angioedema
Brief Title: A Pharmacokinetic, Tolerability and Safety Study of Icatibant in Children and Adolescents With Hereditary Angioedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGT-FIR-086; 2011-003825-81 (EudraCT Number)
Record Dates: First submitted 2011-06-28; First posted 2011-07-01 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: Efficacy; Hereditary angioedema; HAE; Pediatric; Children; Pharmacokinetics; Safety; Firazyr; icatibant
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — icatibant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Icatibant (Experimental): Single dose of icatibant 0.4 mg/kg subcutaneous(SC) up to a maximal dose of 30 mg
  Interventions: Drug: icatibant

INTERVENTIONS:
Drug: icatibant — Single dose of icatibant 0.4 mg/kg subcutaneous(SC) up to a maximal dose of 30 mg
  Other Names: Firazyr

SUMMARY:
HGT-FIR-086 is a multicenter, open-label, non-randomized, single-arm study to evaluate the Pharmacokinetics, tolerability,safety, and efficacy on reproductive hormones, of a single subcutaneous (SC) administration of icatibant in approximately 30 pediatric subjects with Hereditary Angioedema (HAE) during an initial acute attack.

DETAILED DESCRIPTION:
Study HGT-FIR-086 will enroll 30 subjects from 2 to less than 18 years of age, divided into 2 groups: prepubertal and pubertal/postpubertal. At least 10 prepubertal children and at least 20 adolescents (including 10 treated during a HAE attack) must be enrolled in the study.

After a qualifying screening period, the PK, safety/tolerability, and efficacy of treatment with SC icatibant will be evaluated in at least 20 subjects (10 prepubertal and 10 pubertal/postpubertal subjects) who present with cutaneous, abdominal, or laryngeal symptoms of an acute attack of HAE. The PK and safety/tolerability of SC icatibant will be evaluated in at least 10 additional pubertal/postpubertal subjects who meet screening criteria and receive treatment with SC icatibant in the absence of a current acute HAE attack.

The planned duration of active participation for subjects who present with an initial attack of acute HAE will consist of treatment with a single subcutaneous injection of icatibant on Day 1 through follow up at day 90.

After having received initial treatment with icatibant, either during or in the absence of an attack, at least 10 pubertal/postpubertal subjects who subsequently experience an acute HAE attack may continue to receive treatment with icatibant as a single SC administration per attack for a total of 3 eligible icatibant-treated attacks.

The period of active participation in the study for prepubertal subjects will be approximately 90 days, while that for pubertal/postpubertal subjects could be a maximum of approximately 270 or 360 days (3 separate active periods of approximately 90 days for those treated with icatibant during an attack; 4 separate active periods for those treated without an attack), with each active period separated by periods of inactive participation of variable duration.

ELIGIBILITY:
Inclusion Criteria:

1. Two through <18 years of age at the time of first HAE attack.

   * Prepubertal and pubertal/postpubertal subjects experiencing and acute cutaneous, abdominal, or laryngeal HAE attack treated with icatibant as part of this study.
   * Pubertal/postpubertal subjects with HAE who are treated with icatibant, but not during an attack.
2. Documented diagnosis of HAE Type I or II.
3. Informed consent (and subject assent as appropriate) signed by the subject's parent(s)or legal guardian(s).

Exclusion Criteria:

1. Diagnosis of angioedema other than HAE.
2. Participation in another clinical trial that involves the use of any investigational product (drug or device)within 30 days prior to study enrollment or at any time during the study.
3. Any known factor/disease that might interfere with the treatment compliance, study conduct,or result interpretation.
4. Congenital or acquired cardiac anomalies that interfere significantly with cardiac function.
5. Treatment with ACE inhibitors within 7 days prior to treatment.
6. Use of hormonal contraception within the 90 days prior to treatment.
7. Androgen use (eg, stanozolol, danazol, oxandrolone, methyltestosterone, testosterone) within the 90 days prior to treatment.
8. Pregnancy or breastfeeding.
9. A physical condition that interferes with pubertal status determination.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2012-01-27 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (26):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of South Florida, Tampa, Florida
  - Breathe America, Shreveport, Louisiana
  - Institute for Asthma and Allergy, PC, Chevy Chase, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - Oklahoma Institute of Allergy and Asthma Clinical Research, LLC, Oklahoma City, Oklahoma
  - Allergy Asthma Dermatology Research Center, Lake Oswego, Oregon
  - Penn State University, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
- Campbelltown Hospital, Campbelltown, New South Wales, Australia
- Medizinische Universität Graz Hautklinik, Graz, Austria
- McMaster University, Hamilton, Ontario, Canada
- Hospital Infantil Universitario de San Jose, Bogota, Cundinamarca, Colombia
- Germany (3):
  - Klinikum der Johann Wolfgang Goethe University, Frankfurt
  - Johannes-Gutenberg University Clinical Research Center, Mainz
  - HZRM Hämophilie Zentrum Rhein Main GmbH, Walldorf
- Heim Pal Childrens Hospital, Budapest, Hungary
- Israel (3):
  - Bnai Zion Medical Center, Allergy and Immunology Institute, Haifa
  - Tel Aviv Sourasky Medical Center, Pulmonology and Allergy Unit, Tel Aviv
  - Sheba Medical Center Allergy and Immunology Angioedema Center, Tel Litwinsky
- University of Naples Federico II, Dipartimento di Medicina Interna, Naples, Italy
- Spain (2):
  - Unidad de Alergia, Edif. Consultas Externas, Planta Baja HOSPITAL UNIVERSITARIO LA PAZ, Madrid
  - University Hospital, Pediatric Pulmonology and Allergy Unit, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Farkas H, Reshef A, Aberer W, Caballero T, McCarthy L, Hao J, Nothaft W, Schranz J, Bernstein JA, Li HH. Treatment Effect and Safety of Icatibant in Pediatric Patients with Hereditary Angioedema. J Allergy Clin Immunol Pract. 2017 Nov-Dec;5(6):1671-1678.e2. doi: 10.1016/j.jaip.2017.04.010. Epub 2017 Jun 7. PMID 28601641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 27 study centers in the United States, Germany, Israel, Spain, Argentina, Australia, Austria, Canada, Colombia, Hungary, and Italy between 27 January 2012 (first participant first visit) and 12 March 2018 (last participant last visit).
Pre-assignment Details: A total of 32 participants were enrolled and received treatment.
Groups:
- Prepubertal: Participants received a single subcutaneous (SC) injection of 0.4 milligram per kilogram (mg/kg) icatibant (up to a maximal dose of 30 mg) in the abdominal region.
- Pubertal/Postpubertal: Participants received a SC injection of 0.4 mg/kg icatibant (up to a maximal dose of 30 mg) in the abdominal region and participants after receiving initial treatment with icatibant, who subsequently experienced an acute hereditary angioedema (HAE) attack continued to receive treatment with icatibant as a single SC administration per attack for a total of 3 eligible icatibant exposures.
Period: Initial Icatibant Exposure
Arm/Group | Prepubertal | Pubertal/Postpubertal
Started | 11 | 21
Completed | 11 | 9
Not Completed | 0 | 12
Not completed — Withdrawal by Subject | 0 | 9
Not completed — Lack of adherence and poor compliance | 0 | 3
Period: Icatibant Exposure 2
Arm/Group | Prepubertal | Pubertal/Postpubertal
Started | 0 | 9
Completed | 0 | 9
Not Completed | 0 | 0
Period: Icatibant Exposure 3
Arm/Group | Prepubertal | Pubertal/Postpubertal
Started | 0 | 9
Completed | 0 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population consisted of participants who were treated with icatibant at least once during the study.
Groups:
- Prepubertal: Participants received a single SC injection of 0.4 mg/kg icatibant (up to a maximal dose of 30 mg) in the abdominal region.
- Total: Total of all reporting groups
Arm/Group | Prepubertal | Pubertal/Postpubertal | Total
Number analyzed (Participants) | 11 | 21 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.6 (2.97) | 14.3 (1.66) | 12.3 (3.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 6 | 13 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 10 | 19 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 20 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Peak Concentration (Tmax) of a Single Subcutaneous (SC) Dose of Icatibant
Description: Time to peak concentration (Tmax) of a single SC dose of icatibant was reported.
Time Frame: Pre-dose; 0.25, 0.5, 0.75, 1, 2, 4 and 6 hours post-dose on Day 1
Population: Pharmacokinetic (PK) population consisted of participants who were treated with icatibant and had sufficient icatibant plasma concentration-time measurements to derive primary PK parameters. Here the number of participants analyzed signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Hour (h)
Groups:
- Pubertal/Postpubertal: With Acute Attack: Participants with acute attack received a SC injection of 0.4 mg/kg icatibant (up to a maximal dose of 30 mg) in the abdominal region.
- Pubertal/Postpubertal: Without Acute Attack: Participants without acute attack received a SC injection of 0.4 mg/kg icatibant (up to a maximal dose of 30 mg) in the abdominal region.
Arm/Group | Prepubertal | Pubertal/Postpubertal: With Acute Attack | Pubertal/Postpubertal: Without Acute Attack
Number analyzed (Participants) | 9 | 11 | 10
Hour (h) | 0.42 (0.13) | 0.55 (0.19) | 0.57 (0.17)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of a Single Subcutaneous (SC) Dose of Icatibant
Description: Maximum plasma concentration (Cmax) of a single SC dose of icatibant was reported.
Time Frame: Pre-dose; 0.25, 0.5, 0.75, 1, 2, 4 and 6 hours post-dose on Day 1
Population: The PK population consisted of participants who were treated with icatibant and had sufficient icatibant plasma concentration-time measurements to derive primary PK parameters. Here the number of participants analyzed signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Prepubertal | Pubertal/Postpubertal: With Acute Attack | Pubertal/Postpubertal: Without Acute Attack
Number analyzed (Participants) | 9 | 11 | 10
Nanogram per milliliter (ng/mL) | 659 (158) | 805 (125) | 761 (133)

3. Primary Outcome: Total Plasma Clearance (CL/F) of a Single Subcutaneous (SC) Dose of Icatibant
Description: Total plasma clearance (CL/F) of a single SC dose of icatibant was reported.
Time Frame: Pre-dose; 0.25, 0.5, 0.75, 1, 2, 4 and 6 hours post-dose on Day 1
Population: The PK population consisted of participants who were treated with icatibant and had sufficient icatibant plasma concentration time measurements to derive primary PK parameters. Here the number of participants analyzed signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Milliliters per minute (mL/min)
Arm/Group | Prepubertal | Pubertal/Postpubertal: With Acute Attack | Pubertal/Postpubertal: Without Acute Attack
Number analyzed (Participants) | 6 | 11 | 10
Milliliters per minute (mL/min) | 10.8 (4.63) | 13.1 (3.42) | 19.3 (4.84)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 4 Hours Post-dose (AUC0-4) of a Single Subcutaneous (SC) Dose of Icatibant
Description: Area under the plasma concentration-time curve from time zero to 4 hours post-dose (AUC0-4) of a single SC dose of icatibant was reported.
Time Frame: Pre-dose; 0.25, 0.5, 0.75, 1, 2, and 4 hours post-dose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Prepubertal | Pubertal/Postpubertal: With Acute Attack | Pubertal/Postpubertal: Without Acute Attack
Number analyzed (Participants) | 9 | 11 | 10
Hour*nanogram per milliliter (h*ng/mL) | 1241 (319) | 1448 (304) | 1335 (211)

5. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 6 Hours Post-dose (AUC0-t) of a Single Subcutaneous (SC) Dose of Icatibant
Description: Area under the plasma concentration-time curve from time zero to 6 hours post-dose (AUC0-t) of a single SC dose of icatibant was reported.
Time Frame: Pre-dose; 0.25, 0.5, 0.75, 1, 2, 4 and 6 hours post-dose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Prepubertal | Pubertal/Postpubertal: With Acute Attack | Pubertal/Postpubertal: Without Acute Attack
Number analyzed (Participants) | 9 | 11 | 10
h*ng/mL | 1289 (325) | 1573 (372) | 1398 (225)

6. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of a Single Subcutaneous (SC) Dose of Icatibant
Description: Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of a single SC dose of icatibant was reported.
Time Frame: Pre-dose; 0.25, 0.5, 0.75, 1, 2, 4 and 6 hours post-dose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Prepubertal | Pubertal/Postpubertal: With Acute Attack | Pubertal/Postpubertal: Without Acute Attack
Number analyzed (Participants) | 6 | 11 | 10
h*ng/mL | 1243 (244) | 1710 (569) | 1416 (229)

7. Primary Outcome: Volume of Distribution (Vz/F) of a Single Subcutaneous (SC) Dose of Icatibant
Description: Volume of distribution (Vz/F) of a single SC dose of icatibant was reported.
Time Frame: Pre-dose; 0.25, 0.5, 0.75, 1, 2, 4 and 6 hours post-dose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Prepubertal | Pubertal/Postpubertal: With Acute Attack | Pubertal/Postpubertal: Without Acute Attack
Number analyzed (Participants) | 6 | 11 | 10
Liters (L) | 12.5 (5.28) | 23.5 (13.9) | 25.4 (8.87)

8. Primary Outcome: Elimination Half-life (t1/2) of a Single Subcutaneous (SC) Dose of Icatibant
Description: Elimination half-life (t1/2) of a single SC dose of icatibant was reported.
Time Frame: Pre-dose; 0.25, 0.5, 0.75, 1, 2, 4 and 6 hours post-dose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Prepubertal | Pubertal/Postpubertal: With Acute Attack | Pubertal/Postpubertal: Without Acute Attack
Number analyzed (Participants) | 6 | 11 | 10
h | 0.80 (0.04) | 1.34 (0.96) | 0.90 (0.10)

9. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs included pulse rate, blood pressure, respiration rate, and temperature. The number of participants who reported clinically significant changes in vital signs were reported.
Time Frame: Pre-dose up to 97 days post-dose
Population: Safety population consisted of participants who were treated with icatibant at least once during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Prepubertal | Pubertal/Postpubertal
Number analyzed (Participants) | 11 | 21
Participants | 0 | 0

10. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiograms (ECGs)
Description: A standard 12-lead ECG was performed after 10 minutes at rest when the participant was seated or supine following treatment. The number of participants who reported clinically significant changes in ECGs were reported.
Time Frame: 6 - 8 hours post-dose on Day 1
Population: Safety population consisted of participants who were treated with icatibant at least once during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Prepubertal | Pubertal/Postpubertal
Number analyzed (Participants) | 11 | 21
Participants | 0 | 0

11. Primary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Evaluations
Description: Clinical laboratory evaluations included clinical chemistry (including liver function tests), hematology, urinalysis. The number of participants who reported clinically significant changes in clinical laboratory evaluations were reported.
Time Frame: Pre-dose up to 97 days post-dose
Population: Safety population consisted of participants who were treated with icatibant at least once during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Prepubertal | Pubertal/Postpubertal
Number analyzed (Participants) | 11 | 21
Participants | 0 | 0

12. Primary Outcome: Number of Participants Who Reported Presence of Anti-icatibant Antibodies
Description: The number of participants who reported anti-icatibant antibodies were reported.
Time Frame: Pre-dose up to 97 days post-dose
Population: Safety population consisted of participants who were treated with icatibant at least once during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Prepubertal | Pubertal/Postpubertal
Number analyzed (Participants) | 11 | 21
Participants | 0 | 0

13. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in a clinical study, whether or not considered investigational product related.
Time Frame: From the start of study drug administration up to 97 days post-dose
Population: Safety population consisted of participants who were treated with icatibant at least once during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Prepubertal | Pubertal/Postpubertal
Number analyzed (Participants) | 11 | 21
Participants | 2 | 11

14. Primary Outcome: Number of Participants Who Reported Injection Site Reactions (ISR) for Icatibant Exposure Number 1
Description: The number of participants with injection site reactions (erythema, swelling, burning sensation, itching/pruritus, warm sensation, cutaneous pain, or other) that occured after initial icatibant administration was reported.
Time Frame: 1 h post-dose on Day 1 up to 9 days post-dose
Population: Safety population consisted of participants who were treated with icatibant at least once during the study. Here the number of participants analyzed signifies participants who were evaluable for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Prepubertal | Pubertal/Postpubertal
Number analyzed (Participants) | 11 | 21
Participants
  Any Reaction | 9 | 20
  Any Severe Reaction | 0 | 2

15. Primary Outcome: Number of Participants Who Reported Injection Site Reactions (ISR) for Icatibant Exposure Number 2 and 3
Description: The number of participants with injection site reactions (erythema, swelling, burning sensation, itching/pruritus, warm sensation, cutaneous pain, or other) that occurred after subsequent icatibant administration by study-site personnel (health care practitioner [HCP] administration) or by caregiver/self (caregiver administration) was reported. In the below table, E-2 refers to icatibant exposure 2 and E-3 refers to icatibant exposure 3.
Time Frame: 1 h post-dose up to 9 days post-dose
Population: Safety population consisted of participants who were treated with icatibant at least once during the study. Here the number of participants analyzed signifies participants who received subsequent icatibant exposures 2 and 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Pubertal/Postpubertal
Number analyzed (Participants) | 9
Participants
  E-2: HCP Administration: Any Reaction | 1
  E-2: HCP Administration: Any Severe Reaction | 0
  E-2: Caregiver Administration: Any Reaction | 8
  E-2: Caregiver Administration: Any Severe Reaction | 3
  E-3: HCP Administration: Any Reaction | 1
  E-3: HCP Administration: Any Severe Reaction | 0
  E-3: Caregiver Administration: Any Reaction | 7
  E-3: Caregiver Administration: Any Severe Reaction | 1

16. Primary Outcome: Number of Participants With Clinically Significant Changes in Reproductive Hormones
Description: Reproductive hormone levels of follicle-stimulating hormone (FSH), luteinizing hormone (LH), estradiol, and progesterone in females, and FSH, LH, and testosterone in males were measured. The number of participants with clinically significant changes in reproductive hormones was reported.
Time Frame: Pre-dose up to 97 days post-dose
Population: Safety population consisted of participants who were treated with icatibant at least once during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Prepubertal | Pubertal/Postpubertal
Number analyzed (Participants) | 11 | 21
Participants | 0 | 0

17. Secondary Outcome: Time to Onset of Symptom Relief (TOSR) for Composite Investigator-Assessed Symptom Scores for Icatibant Exposure Number 1
Description: The TOSR was defined as the duration of time in hours from study drug administration to the earliest time post-treatment at which there was at least a 20 percent (%) improvement in the average post-treatment symptom score with no worsening of any single component score for the initial icatibant exposure. The investigator used a symptom score to assess the severities of symptoms of acute cutaneous, abdominal, and laryngeal attacks of hereditary angioedema (HAE) using the following 5-point scale: 0=none (absence of symptoms), 1=mild (no to mild interference with daily activities), 2=moderate (moderate interference with daily activities), 3=severe (severe interference with daily activities) and 4=very severe (very severe interference with daily activities). TOSR for participants who received initial icatibant administration was reported.
Time Frame: From start of study drug administration up to 8.5 hours post-dose
Population: Efficacy population consisted of participants who were treated with icatibant for their first and any additional attacks during the study. Here the number of participants analyzed signifies participants who were evaluable for this measure.
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Prepubertal | Pubertal/Postpubertal
Number analyzed (Participants) | 11 | 11
h | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]

18. Secondary Outcome: Time to Onset of Symptom Relief (TOSR) for Composite Investigator-Assessed Symptom Scores for Icatibant Exposure Number 2 and 3
Description: The TOSR was defined as the duration of time in hours from study drug administration to the earliest time post-treatment at which there was at least a 20% improvement in the composite (or average) post-treatment symptom score with no worsening of any single component score. The investigator used a symptom score to assess the severities of symptoms of acute cutaneous, abdominal, and laryngeal attacks of HAE using the following 5-point scale: 0=none (absence of symptoms), 1=mild (no to mild interference with daily activities), 2=moderate (moderate interference with daily activities), 3=severe (severe interference with daily activities) and 4=very severe (very severe interference with daily activities). TOSR for participants who received subsequent icatibant administration by HCP administration or by caregiver/ self-administration was reported.
Time Frame: From start of study drug administration up to 12 hours post-dose
Population: Efficacy population consisted of participants who were treated with icatibant for their first and any additional attacks during the study. Here the number of participants analyzed signifies participants who received subsequent icatibant exposures 2 and 3.
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Pubertal/Postpubertal
Number analyzed (Participants) | 9
h
  Icatibant Exposure-2: HCP Administration: number analyzed (Participants) | 1
  Icatibant Exposure-2: HCP Administration | 4.0 [NA to NA] — Percentage confidence interval (%CI) was not calculated due to less number of participants.
  Icatibant Exposure-2: Caregiver Administration: number analyzed (Participants) | 8
  Icatibant Exposure-2: Caregiver Administration | 1.0 [1.0 to 2.3]
  Icatibant Exposure-3: HCP Administration: number analyzed (Participants) | 1
  Icatibant Exposure-3: HCP Administration | 1.0 [NA to NA] — %CI was not calculated due to less number of participants.
  Icatibant Exposure-3:Caregiver Administration: number analyzed (Participants) | 7
  Icatibant Exposure-3:Caregiver Administration | 1.1 [1.0 to 3.0]

19. Secondary Outcome: Time to Onset of Symptom Relief (TOSR) for Faces Pain Scale-Revised (FPS-R) Scores for Icatibant Exposure Number 1
Description: The TOSR was defined as the earliest time at which the post-treatment score improved by at least one level. Participants of 4 years age and older self-assessed their HAE-related pain using the FPS-R instrument. FPS-R is a self-reported measure used to assess the intensity of children's pain and it is scored using a 0 to 10 scale (0=no pain to 10=very much pain). TOSR for participants who received initial icatibant administration was reported.
Time Frame: From start of study drug administration up to 52 hours post-dose
Population: Efficacy population consisted of participants who were treated with icatibant for their first and any additional attacks during the study. Here the number of participants analyzed signifies participants with FPS-R data.
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Prepubertal | Pubertal/Postpubertal
Number analyzed (Participants) | 6 | 9
h | 0.9 [0.8 to 1.0] | 1.0 [0.6 to 1.0]

20. Secondary Outcome: Time to Onset of Symptom Relief (TOSR) for Faces Pain Scale-Revised (FPS-R) Scores for Icatibant Exposure Number 2 and 3
Description: The TOSR was defined as the earliest time at which the post-treatment score improved by at least one level. Participants of 4 years age and older self-assessed their HAE-related pain using the FPS-R instrument. FPS-R is a self-reported measure used to assess the intensity of children's pain and it is scored using a 0 to 10 scale (0=no pain to 10=very much pain). TOSR for participants who received subsequent icatibant administration by HCP administration or by caregiver/ self-administration was reported.
Time Frame: From start of study drug administration up to 28 hours post-dose
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Pubertal/Postpubertal
Number analyzed (Participants) | 9
h
  Icatibant Exposure-2: HCP Administration: number analyzed (Participants) | 1
  Icatibant Exposure-2: HCP Administration | 3.0 [NA to NA] — %CI was not calculated due to less number of participants.
  Icatibant Exposure-2: Caregiver Administration: number analyzed (Participants) | 7
  Icatibant Exposure-2: Caregiver Administration | 1.0 [1.0 to 1.2]
  Icatibant Exposure-3: HCP Administration: number analyzed (Participants) | 1
  Icatibant Exposure-3: HCP Administration | 1.0 [NA to NA] — %CI was not calculated due to less number of participants.
  Icatibant Exposure-3:Caregiver Administration: number analyzed (Participants) | 7
  Icatibant Exposure-3:Caregiver Administration | 1.1 [1.0 to 1.2]

21. Secondary Outcome: Time to Onset of Symptom Relief (TOSR) for Faces, Legs, Activity, Cry, and Consolability (FLACC) Scores
Description: The TOSR was defined as the earliest time at which a 20% improvement was seen in the total post-treatment score. Participants of 4 years age and younger underwent investigator assessment of HAE-related pain (cutaneous, abdominal, and laryngeal) using the FLACC comportmental pain scale. Each of the 5 categories was scored from 0 to 2. Face(F): 0 (no particular expression/smile) - 2 (frequent to constant frown clenched jaw quivering chin); Legs(L): 0 (normal position/relaxed) - 2 (kicking/legs drawn up); Activity(A): 0 (lying quietly, normal position, moves easily) - 2 (arched rigid/jerking); Cry(C): 0 (No cry [awake/asleep]) - 2 (crying steadily/screams/sobs or frequent complaints); Consolability(C): 0 (content/relaxed) - 2 (difficult to console/comfort), resulting in a total score between 0 and 10.
Time Frame: From start of study drug administration up to 8.5 hours post-dose
Population: Efficacy population consisted of participants who were treated with icatibant for their first and any additional attacks during the study. Here the number of participants analyzed signifies participants of 4 years and younger with FLACC data.
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Prepubertal
Number analyzed (Participants) | 1
h | 1.0 [NA to NA] — %CI was not calculated due to less number of participants.

22. Secondary Outcome: Time to Minimum Symptoms for Composite Investigator-Assessed Symptom Scores for Icatibant Exposure Number 1
Description: Time to minimum symptom was defined as the duration of time in hours from study drug administration to the earliest time post-treatment at which all symptoms were either mild or absent for the investigator-reported symptom score. The investigator used a symptom score to assess the severities of symptoms of acute cutaneous, abdominal, and laryngeal attacks of HAE using the following 5-point scale: 0=none (absence of symptoms), 1=mild (no to mild interference with daily activities), 2=moderate (moderate interference with daily activities), 3=severe (severe interference with daily activities) and 4=very severe (very severe interference with daily activities). Time to minimum symptom for participants who received initial icatibant administration was reported.
Time Frame: From start of study drug administration up to 8.5 hours post-dose
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Prepubertal | Pubertal/Postpubertal
Number analyzed (Participants) | 11 | 10
h | 1.9 [1.0 to 2.0] | 1.0 [1.0 to 2.0]

23. Secondary Outcome: Time to Minimum Symptoms for Composite Investigator-Assessed Symptom Scores for Icatibant Exposure Number 2 and 3
Description: Time to minimum symptom was defined as the duration of time in hours from study drug administration to the earliest time post-treatment at which all symptoms were either mild or absent for the investigator-reported symptom score. The investigator used a symptom score to assess the severities of symptoms of acute cutaneous, abdominal, and laryngeal attacks of HAE using the following 5-point scale: 0=none (absence of symptoms), 1=mild (no to mild interference with daily activities), 2=moderate (moderate interference with daily activities), 3=severe (severe interference with daily activities) and 4=very severe (very severe interference with daily activities). Time to minimum symptom for participants who received subsequent icatibant administration by HCP administration or by caregiver/ self-administration was reported.
Time Frame: From start of study drug administration up to 12 hours post-dose
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Pubertal/Postpubertal
Number analyzed (Participants) | 9
h
  Icatibant Exposure-2: HCP Administration: number analyzed (Participants) | 0
  Icatibant Exposure-2: Caregiver Administration: number analyzed (Participants) | 7
  Icatibant Exposure-2: Caregiver Administration | 1.2 [1.0 to 2.0]
  Icatibant Exposure-3: HCP Administration: number analyzed (Participants) | 0
  Icatibant Exposure-3: Caregiver Administration: number analyzed (Participants) | 7
  Icatibant Exposure-3: Caregiver Administration | 2.2 [1.0 to NA] — The data was not calculated due to analysis method limitation.

24. Secondary Outcome: Time to Minimum Symptom for Faces Pain Scale-Revised (FPS-R) Scores for Icatibant Exposure Number 1
Description: Time to minimum symptoms was defined as the duration of time in hours from study drug administration to the earliest time at which post-treatment score improved to zero (or no pain). Participants of 4 years of age and older self-assessed their HAE-related pain using the FPS-R instrument. FPS-R is a self-reported measure used to assess the intensity of children's pain and it is scored using a 0 to 10 scale (0=no pain to 10=very much pain). Time to minimum symptom for participants who received initial icatibant administration was reported.
Time Frame: From start of study drug administration up to 52 hours post-dose
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Prepubertal | Pubertal/Postpubertal
Number analyzed (Participants) | 6 | 11
h | 2.4 [1.9 to 5.3] | 3.8 [1.0 to 6.8]

25. Secondary Outcome: Time to Minimum Symptom for Faces Pain Scale-Revised (FPS-R) Scores for Icatibant Exposure Number 2 and 3
Description: Time to minimum symptoms was defined as the duration of time in hours from study drug administration to the earliest time at which post-treatment score improved to zero (or no pain). Participants of 4 years of age and older self-assessed their HAE-related pain using the FPS-R instrument. FPS-R is a self-reported measure used to assess the intensity of children's pain and it is scored using a 0 to 10 scale (0=no pain to 10=very much pain). Time to minimum symptom for participants who received subsequent icatibant administration by HCP administration or by caregiver/ self-administration was reported.
Time Frame: From start of study drug administration up to 28 hours post-dose
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Pubertal/Postpubertal
Number analyzed (Participants) | 9
h
  Icatibant Exposure-2: HCP Administration: number analyzed (Participants) | 1
  Icatibant Exposure-2: HCP Administration | 3.0 [NA to NA] — The %CI was not calculated due to less number of participants.
  Icatibant Exposure-2: Caregiver Administration: number analyzed (Participants) | 7
  Icatibant Exposure-2: Caregiver Administration | 2.1 [1.0 to 4.0]
  Icatibant Exposure-3: HCP Administration: number analyzed (Participants) | 1
  Icatibant Exposure-3: HCP Administration | 5.8 [NA to NA] — The %CI was not calculated due to less number of participants.
  Icatibant Exposure-3:Caregiver Administration: number analyzed (Participants) | 7
  Icatibant Exposure-3:Caregiver Administration | 24.0 [3.8 to 24.2]

26. Secondary Outcome: Time to Minimum Symptom for Faces, Legs, Activity, Cry, and Consolability (FLACC) Scores
Description: Time to minimum symptoms was defined as the duration of time in hours from study drug administration to the earliest time at which the total post-treatment score improved to zero. Participants of 4 years age and younger underwent investigator assessment of HAE-related pain (cutaneous, abdominal, and laryngeal) using the FLACC comportmental pain scale. Each of the 5 categories was scored from 0 to 2. (F) Face: 0 (no particular expression/smile) - 2 (frequent to constant frown clenched jaw quivering chin); (L) Legs: 0 (normal position/relaxed) - 2 (kicking/legs drawn up); (A) Activity: 0 (lying quietly, normal position, moves easily) - 2 (arched rigid/jerking); (C) Cry: 0 (No cry [awake/asleep]) - 2 (crying steadily/screams/sobs or frequent complaints); (C) Consolability: 0 (content/relaxed) - 2 (difficult to console/comfort), resulting in a total score between 0 and 10.
Time Frame: From start of study drug administration up to 8.5 hours post-dose
Population: Participants from efficacy population with FLACC data.
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Prepubertal
Number analyzed (Participants) | 1
h | 1.0 [NA to NA] — The %CI was not calculated due to less number of participants.

27. Secondary Outcome: Time to Use of Rescue Medication for the Treatment of Symptoms of the Hereditary Angioedema (HAE) Attack Following Study Drug Administration
Description: Rescue medication was any medication used after the administration of icatibant which, in the opinion of the investigator, was immediately necessary to alleviate acute symptoms which are judged by the investigator as resultant from the current HAE attack. Time to first use of rescue medication prior to the onset of symptom relief was calculated from the time of study drug administration to the first use of rescue medication prior to the onset of symptom relief. This analysis was not performed since as per protocol, "This analysis will only be performed if there are at least 5 participants for a given attack who used rescue medication prior to attaining symptom relief".
Time Frame: From the start of study drug administration up to 52 hours post-dose
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Prepubertal | Pubertal/Postpubertal
Number analyzed (Participants) | 11 | 11
h | NA [NA to NA] — This analysis was planned to be performed if there were at least 5 participants for a given attack who used rescue medication prior to attaining symptom relief. | NA [NA to NA] — This analysis was planned to be performed if there were at least 5 participants for a given attack who used rescue medication prior to attaining symptom relief.

28. Secondary Outcome: Number of Participants With Worsened Intensity of Clinical Hereditary Angioedema (HAE) Symptoms Between 2 and 4 Hours After Treatment With Icatibant Exposure Number 1
Description: The investigator used a symptom score to assess the severities of symptoms of acute cutaneous, abdominal, and laryngeal attacks of HAE using the following 5- point scale: 0=none (absence of symptoms), 1=mild (no to mild interference with daily activities), 2=moderate (moderate interference with daily activities), 3=severe (severe interference with daily activities) and 4=very severe (very severe interference with daily activities). The number of participants with a worsened severity of HAE symptoms at 4 hours post-dose from 2 hours postdose were reported.
Time Frame: From 2 hours post-dose to 4 hours post-dose
Population: Efficacy population consisted of participants who were treated with icatibant for their first and any additional attacks during the study. Here the number of participants analyzed signifies participants who evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Prepubertal | Pubertal/Postpubertal
Number analyzed (Participants) | 11 | 11
Participants
  Abdominal Tenderness | 0 | 1
  Nausea | 0 | 0
  Vomiting | 0 | 0
  Diarrhea | 0 | 0
  Skin Pain | 0 | 0
  Erythema | 0 | 0
  Skin Irritation | 0 | 0
  Skin Swelling | 0 | 0

29. Secondary Outcome: Number of Participants With Worsened Intensity of Clinical Hereditary Angioedema (HAE) Symptoms Between 2 and 4 Hours After Treatment With Icatibant Exposure Number 2 and 3
Description: The investigator used a symptom score to assess the severities of symptoms of acute cutaneous, abdominal, and laryngeal attacks of HAE using the following 5- point scale: 0=none (absence of symptoms), 1=mild (no to mild interference with daily activities), 2=moderate (moderate interference with daily activities), 3=severe (severe interference with daily activities) and 4=very severe (very severe interference with daily activities). The number of participants with a worsened severity of HAE symptoms at 4 hours post-dose from 2 hours post-dose were reported.
Time Frame: From 2 hours post-dose to 4 hours post-dose
Population: Efficacy population consisted of participants who were treated with icatibant for their first and any additional attacks during the study. The number of participants analyzed signifies participants evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Pubertal/Postpubertal
Number analyzed (Participants) | 9
Participants
  E-2: HCPA: Abdominal Tenderness: number analyzed (Participants) | 1
  E-2: HCPA: Abdominal Tenderness | 0
  E-2:CA: Abdominal Tenderness: number analyzed (Participants) | 8
  E-2:CA: Abdominal Tenderness | 0
  E-2: HCPA: Nausea: number analyzed (Participants) | 1
  E-2: HCPA: Nausea | 0
  E-2: CA: Nausea: number analyzed (Participants) | 8
  E-2: CA: Nausea | 0
  E-2:HCPA: Vomiting: number analyzed (Participants) | 1
  E-2:HCPA: Vomiting | 0
  E-2: CA: Vomiting: number analyzed (Participants) | 8
  E-2: CA: Vomiting | 0
  E-2: HCPA: Diarrhea: number analyzed (Participants) | 1
  E-2: HCPA: Diarrhea | 0
  E-2: CA: Diarrhea: number analyzed (Participants) | 8
  E-2: CA: Diarrhea | 0
  E-2: HCPA: Skin Pain: number analyzed (Participants) | 1
  E-2: HCPA: Skin Pain | 0
  E-2: CA: Skin Pain: number analyzed (Participants) | 8
  E-2: CA: Skin Pain | 0
  E-2: HCPA: Erythema: number analyzed (Participants) | 1
  E-2: HCPA: Erythema | 0
  E-2: CA: Erythema: number analyzed (Participants) | 8
  E-2: CA: Erythema | 0
  E-2: HCPA: Skin Irritation: number analyzed (Participants) | 1
  E-2: HCPA: Skin Irritation | 0
  E-2: CA: Skin Irritation: number analyzed (Participants) | 8
  E-2: CA: Skin Irritation | 0
  E-2: HCPA: Skin Swelling: number analyzed (Participants) | 1
  E-2: HCPA: Skin Swelling | 0
  E-2: CA: Skin Swelling: number analyzed (Participants) | 8
  E-2: CA: Skin Swelling | 0
  E-2: HCPA: Dysphagia: number analyzed (Participants) | 1
  E-2: HCPA: Dysphagia | 0
  E-2: CA: Dysphagia: number analyzed (Participants) | 8
  E-2: CA: Dysphagia | 0
  E-2: HCPA: Voice Change: number analyzed (Participants) | 1
  E-2: HCPA: Voice Change | 0
  E-2: CA: Voice Change: number analyzed (Participants) | 8
  E-2: CA: Voice Change | 0
  E-2: HCPA: Breathing Difficulties: number analyzed (Participants) | 1
  E-2: HCPA: Breathing Difficulties | 0
  E-2: CA: Breathing Difficulties: number analyzed (Participants) | 8
  E-2: CA: Breathing Difficulties | 0
  E-2: HCPA: Stridor: number analyzed (Participants) | 1
  E-2: HCPA: Stridor | 0
  E-2: CA: Stridor: number analyzed (Participants) | 8
  E-2: CA: Stridor | 0
  E-2: HCPA: Asphyxia: number analyzed (Participants) | 1
  E-2: HCPA: Asphyxia | 0
  E-2:CA: Asphyxia: number analyzed (Participants) | 8
  E-2:CA: Asphyxia | 0
  E-3: HCPA: Abdominal Tenderness: number analyzed (Participants) | 1
  E-3: HCPA: Abdominal Tenderness | 0
  E-3: CA: Abdominal Tenderness: number analyzed (Participants) | 8
  E-3: CA: Abdominal Tenderness | 1
  E-3: HCPA: Nausea: number analyzed (Participants) | 1
  E-3: HCPA: Nausea | 0
  E-3: CA: Nausea: number analyzed (Participants) | 8
  E-3: CA: Nausea | 0
  E-3: HCPA: Vomiting: number analyzed (Participants) | 1
  E-3: HCPA: Vomiting | 0
  E-3: CA: Vomiting: number analyzed (Participants) | 8
  E-3: CA: Vomiting | 0
  E-3: HCPA: Diarrhea: number analyzed (Participants) | 1
  E-3: HCPA: Diarrhea | 0
  E-3: CA: Diarrhea: number analyzed (Participants) | 8
  E-3: CA: Diarrhea | 1
  E-3: HCPA: Skin Pain: number analyzed (Participants) | 1
  E-3: HCPA: Skin Pain | 0
  E-3: CA: Skin Pain: number analyzed (Participants) | 8
  E-3: CA: Skin Pain | 0
  E-3: HCPA: Erythema: number analyzed (Participants) | 1
  E-3: HCPA: Erythema | 0
  E-3: CA: Erythema: number analyzed (Participants) | 8
  E-3: CA: Erythema | 0
  E-3: HCPA: Skin Irritation: number analyzed (Participants) | 1
  E-3: HCPA: Skin Irritation | 0
  E-3: CA: Skin Irritation: number analyzed (Participants) | 8
  E-3: CA: Skin Irritation | 0
  E-3: HCPA: Skin Swelling: number analyzed (Participants) | 1
  E-3: HCPA: Skin Swelling | 0
  E-3: CA: Skin Swelling: number analyzed (Participants) | 8
  E-3: CA: Skin Swelling | 0
  E-3: HCPA: Dysphagia: number analyzed (Participants) | 1
  E-3: HCPA: Dysphagia | 0
  E-3: CA: Dysphagia: number analyzed (Participants) | 8
  E-3: CA: Dysphagia | 0
  E-3: HCPA: Voice Change: number analyzed (Participants) | 1
  E-3: HCPA: Voice Change | 0
  E-3: CA: Voice Change: number analyzed (Participants) | 8
  E-3: CA: Voice Change | 0
  E-3: HCPA: Breathing Difficulties: number analyzed (Participants) | 1
  E-3: HCPA: Breathing Difficulties | 0
  E-3: CA: Breathing Difficulties: number analyzed (Participants) | 8
  E-3: CA: Breathing Difficulties | 0
  E-3: HCPA: Stridor: number analyzed (Participants) | 1
  E-3: HCPA: Stridor | 0
  E-3: CA: Stridor: number analyzed (Participants) | 8
  E-3: CA: Stridor | 0
  E-3: HCPA: Asphyxia: number analyzed (Participants) | 1
  E-3: HCPA: Asphyxia | 0
  E-3: CA: Asphyxia: number analyzed (Participants) | 8
  E-3: CA: Asphyxia | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 187 days
Groups:
- Pubertal/Post-pubertal: Participants received a SC injection of 0.4 mg/kg icatibant (up to a maximal dose of 30 mg) in the abdominal region and participants after receiving initial treatment with icatibant, who subsequently experienced an acute hereditary angioedema (HAE) attack continued to receive treatment with icatibant as a single SC administration per attack for a total of 3 eligible icatibant exposures.
- Overall: Participants received a single subcutaneous(SC) injection of 0.4 mg/kg icatibant (up to a maximal dose of 30 mg) in the abdominal region. Pubertal/postpubertal participants after receiving initial treatment with icatibant, who subsequently experienced an acute hereditary angioedema (HAE) attack continued to receive treatment with icatibant as a single SC administration per attack for a total of 3 eligible icatibant exposures.
Arm/Group | Prepubertal | Pubertal/Post-pubertal | Overall
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/21 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/21 | 0/32
Other Adverse Events (participants affected / at risk) | 4/11 | 8/21 | 12/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prepubertal (N=11) | Pubertal/Post-pubertal (N=21) | Overall (N=32)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (5) | 2 (5)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 2 (9) | 2 (9)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (4) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (3) | 3 (4)
Epiphyseal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Nitrite urine present (Investigations) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 1 (1) | 2 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (6):
  • Study Protocol: Protocol Original (2011-06-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT01386658/Prot_000.pdf
  • Study Protocol: Protocol Amendment 1 (2011-08-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT01386658/Prot_001.pdf
  • Study Protocol: Protocol Amendment 2 (2012-03-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT01386658/Prot_002.pdf
  • Study Protocol: Protocol Amendment 3 (2013-06-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT01386658/Prot_003.pdf
  • Study Protocol: Protocol Amendment 4 (2016-03-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT01386658/Prot_004.pdf
  • Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT01386658/SAP_005.pdf